CLINICAL TRIAL: NCT03046589
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Oral Dose, Safety, Tolerability, Pharmacodynamic, and Pharmacokinetic Study of DP13 in Healthy Male Subjects
Brief Title: DP13 SAD & MAD in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Damian Pharma AG (Industry)
Collaborators: Covance (Industry); Foundation for Therapeutic Research, Lausanne (Unknown); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DP13C101
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2017-07

CONDITIONS: Safety and Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment Period 1 (Experimental): DP13 capsules (dose level 1 ) and placebo capsules
  Interventions: Drug: DP13; Drug: placebo
- Treatment Period 2 (Experimental): DP13 capsules (dose level 2) and placebo capsules
  Interventions: Drug: DP13; Drug: placebo
- Treatment Period 3 (Experimental): DP13 capsules (dose level 3) and placebo capsules
  Interventions: Drug: DP13; Drug: placebo
- Treatment Period 4 (Experimental): DP13 capsules (dose level 4) and placebo capsules
  Interventions: Drug: DP13; Drug: placebo
- Treatment Period 5 (Experimental): DP13 capsules (dose level 5) and placebo capsules
  Interventions: Drug: DP13; Drug: placebo
- Treatment Period 6 (Experimental): DP13 capsules (dose level 6) and placebo capsules
  Interventions: Drug: DP13; Drug: placebo

INTERVENTIONS:
Drug: DP13 — dose escalation
Drug: placebo — control to dose-escalation

SUMMARY:
Primary Objectives:

1. To determine the safety and tolerability of single and multiple oral doses of DP13 in healthy male subjects
2. To assess the pharmacodynamics of single and multiple ascending oral doses as well as dosing regimen of DP13 on suppression of serum aldosterone in healthy male subjects

Secondary Objectives:

1. To determine the single and multiple oral dose pharmacokinetics of DP13 in healthy male subjects
2. To determine the dose-dependent pharmacodynamic selectivity of DP13 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 18.0 and 30.0 kg/m2, inclusive
2. body weight between 60 and 95 kg, inclusive
3. good health as determined by medical history, physical examination, vital signs assessment, 12-lead ECG, clinical laboratory evaluations
4. normal stress response
5. sodium value within the normal laboratory reference range
6. potassium value within the normal laboratory reference range
7. written informed consent

Exclusion Criteria:

1. unwilling to consent or whose partner is unwilling to consent to use a barrier method of contraception
2. blood donation within 3 months prior to screening or plasma donation within 7 days prior to screening or platelet donation within 6 weeks prior to screening
3. consumption of more than 28 units of alcohol per week or significant history of alcoholism or drug/chemical abuse within the last 12 months prior to screening
4. use of tobacco or nicotine-containing products within 3 months
5. use of any of the following within 14 days of first dose: non-prescribed systemic or topical medication; any herbal remedy; any vitamin supplement; any mineral supplement
6. receipt of any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes
7. receipt or intent to receive: any prescribed systemic or topical medication within 14 days of first dose administration
8. an abnormality in heart rate, blood pressure, temperature or respiration rate at screening and prior to first dose that in the opinion of the investigator increases the risk of participating in the study
9. a positive urine drugs of abuse screen
10. an abnormality in the 12-lead ECG at screening and prior to first dose that in the opinion of the investigator increases the risk of participating in the study
11. a medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome
12. participation in another clinical study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (Clinical signs and symptoms incl ECG, vital signs, electrolytes) | Up to 2 weeks after dosing
  Clinical signs and symptoms incl ECG, vital signs, electrolytes
Aldosterone suppression | Up to 48 hours after dosing
  Serum aldosterone concentration

SECONDARY OUTCOMES:
Pharmacokinetics (Plasma DP13 concentration) | up to 48 hours after dosing
  Plasma DP13 concentration
Pharmacodynamic selectivity (Plasma hormone concentrations) | Up to 48 hours after dosing
  Plasma hormone concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MBChB, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulatero P, Groessl M, Vogt B, Schumacher C, Steele RE, Brooks A, Hossack S, Brunner HR. CYP11B2 inhibitor dexfadrostat phosphate suppresses the aldosterone-to-renin ratio, an indicator of sodium retention, in healthy volunteers. Br J Clin Pharmacol. 2023 Aug;89(8):2483-2496. doi: 10.1111/bcp.15713. Epub 2023 Apr 10. PMID 36914591